CLINICAL TRIAL: NCT05892302
Title: A Culturally Tailored Scalable Asthma Intervention for Hispanic Children
Brief Title: A Culturally Tailored Scalable Asthma Intervention for Hispanic Children (Asthma Guardian)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas at Austin (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Elizabeth Matsui, Professor, Departments of Population Health and Pediatrics, University of Texas at Austin
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: STUDY00004576; R34HL159126 (NIH)
Record Dates: First submitted 2023-05-17; First posted 2023-06-07 (Actual); Last update posted 2024-07-01 (Actual); Status verified 2024-06

CONDITIONS: Asthma in Children

STUDY DESIGN:
Masking Description: Only the statistician will be blinded to study group.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Access to Asma Guardian website/app (Active Comparator): Participants who are randomized to the Asma Guardian website at their baseline visit will have access to the website for 6 months starting at baseline. Access will be turned off at 6 months.
  Interventions: Behavioral: Access to Asma Guardian website/app
- No Access to Asma Guardian website/app for 6 months (Other): Note: Participants who are randomized to no access will not receive access during the 6 months of the study; however they will receive 1 month of access after their 6 month study visit but any information gained during this time will not be part of analysis.
  Interventions: Behavioral: Delayed Access to Asma Guardian website/app

INTERVENTIONS:
Behavioral: Access to Asma Guardian website/app — The Asma Guardian intervention application is a culturally-tailored web-platform that includes 3 tool kits. The contents of the tool kits include Asthma Specialty Care, Family Asthma Management, and Home Environmental Intervention.
  Arms: Access to Asma Guardian website/app
Behavioral: Delayed Access to Asma Guardian website/app — Delayed access to the website/app. The Asma Guardian intervention application is a culturally-tailored web-platform that includes 3 tool kits. The contents of the tool kits include Asthma Specialty Care, Family Asthma Management, and Home Environmental Intervention.
  Arms: No Access to Asma Guardian website/app for 6 months

SUMMARY:
This is a two-arm, parallel design, randomized, controlled pilot trial comparing access to Asma Guardián, a culturally tailored multi-component app-based asthma intervention for Hispanic/Latinx school age children with asthma, to usual care.

DETAILED DESCRIPTION:
This is a pilot two-arm, parallel design, randomized, controlled clinical trial that will test a scalable, culturally-tailored, multilayered asthma intervention, Asthma Guardian, designed to reduce asthma morbidity among Mexican American/Hispanic children. This study will inform the planning of a statewide efficacy trial. Asthma Guardian will include three components: (1) support for accessing asthma specialist care, (2) asthma management education and support, and (3) home environment education, access to housing advocacy services, and access to environmental intervention supplies. These components will be accessed by families through a web-based platform, which will include educational materials, a portal for requesting environmental intervention supplies, and access to a virtual community health worker (vCHW), who will facilitate engagement with subspecialty care and housing advocacy services and support asthma self-management. A trained vCHW will communicate with families via telephone and/or video calls. The Investigators will examine Asthma Guardian's effects on clinical outcomes as well as process/fidelity outcomes, including uptake and implementation of the toolkits, education, vCHW support, and environmental intervention supplies. The Investigators propose achieving this goal by randomizing 50 Mexican American/Hispanic children with uncontrolled asthma to either immediate or delayed access (6 months after randomization for one month) to the Asthma Guardian platform. Participants randomized to receive immediate access will be enrolled for 6 months.

A randomization table will be generated by the study statistician and implemented through RedCAP. Using a computer-based algorithm accessed by web-enabled tablet, participants will be randomized 1:1 to the two conditions using a random block size (of 4 or 6) algorithm so that the order of randomization is not predictable by any study team member. The randomization scheme will only be accessible to the data manager. Participants will be given a unique ID number to logon to the website where they can access the vCHW and tool kits.

A participant is considered to have completed the study if he or she has completed the baseline assessment, receive access to intervention application (either at baseline or 6 month mark), and the 6-month follow-up assessments.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of signed and dated informed consent forms.
2. Who has a child who is 5-12 years of age
3. Whose child meets criteria for current persistent asthma defined as either:

   1. On a long-term controller medication for asthma, or
   2. Meet NAEPP guideline requirements for persistent disease:)(35)

      * Asthma symptoms 3 or more days per week over the past 2 weeks OR
      * Nocturnal asthma symptoms at least 3 times in the past month
4. Whose child has had an asthma exacerbation, defined as an oral steroid burst, in the previous 12 months
5. Parent/Caregiver identifies as Mexican American or other Hispanic descent
6. Whose child has clinician diagnosed asthma
7. Access to necessary resources for participating in a technology-based intervention (i.e., computer, smart phone, internet access)
8. Whose child is not currently participating in another asthma study.

The parent/caregiver is the primary study participant, but the child will be asked to complete some surveys at baseline and six months, so an assent will be obtained from the child.

Exclusion Criteria:

* An individual who meets any of the following criteria will be excluded from participation in this study:

  1. Unwilling to provide consent for research activities
  2. Cognitive inability to provide consent
  3. Whose child has evidence of other chronic lung or significant cardiovascular disease
  4. Whose child has a history of intubation for asthma

Ages: 5 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 50 (Estimated)
Dates: Start 2024-03-22 (Actual); Primary Completion 2025-04-01 (Estimated); Study Completion 2025-05-01 (Estimated)

PRIMARY OUTCOMES:
Participant engagement with the Asthma Guardian website/app | 6 months
  Engagement is a composite outcome which is defined as engagement with at least 2 of the 3 toolkits. It will be expressed as the percentage of participants with engagement. Engagement with each of the toolkits is defined as follows:
  (i) Asthma Specialist: at least one documented appointment with an asthma specialist; (ii) Asthma Management: Controller medication prescription fills covering at least 3 months of dosing; (iii) Home environment Toolkit: New deployment of at least some of the available environmental intervention materials, such as air purifiers.

OTHER OUTCOMES:
Asthma Control Test (ACT) | 6 months follow-up visit
  Score range 5-25, higher score indicates better outcome.
Asthma Exacerbation | 6 months
  Defined as an oral steroid burst, measured as the number of bursts taken over the six month follow-up period
Asthma related acute care use | 6 months
  Measured by the number of hospitalizations, ER visits, or Unexpected Doctor visits over the six month follow-up period
Asthma controller medication | 6 month follow-up visit
  Measured by the number of days controller medication was taken in a 2 week period
Asthma controller medication treatment step | 6 month follow-up visit
  controller medication treatment step at the 6 month follow-up visit
Asthma symptoms | 6 month follow-up visit
  number of days of asthma symptoms in the previous 2 weeks
Asthma Specialty Visit | 6 months
  Defined as reporting at least one visit with an asthma specialist during the six month follow-up period
Short adapted Questionnaire to Measure Asthma Knowledge of Parents. | 6 months
  Measured using the Asthma Knowledge Questionnaire, sum of the scores for each question A Likert-type scale of 5 points is used. Items are graded '1', '2', '3', '4', and '5' for 'strongly disagree', 'disagree', 'neither agree, nor disagree', 'agree', and 'strongly agree', respectively.
  Negative items are reverse coded by subtracting the responses values from 5. Missing answers of the asthma knowledge questionnaire scores a '3'. Total score is calculated by the sum of score item responses, ranging from 10 to 50, with higher scores indicating greater knowledge of asthma.
Pharmacy prescription data | 6 months
  Number of asthma controller medication prescription fills over the six month follow-up period
Use of the asthma control test | 6 months
  defined as the number of times the ACT form is downloaded from the app over the six month follow-up period
Request for home environmental supplies | 6 months
  Defined as the number of requests for home environmental supplies in the app over the six month time period
Deployment of home environmental supplies | 6 months
  Defined as report of deployment of any environmental supplies during the six month follow-up visits
Settled Dust allergen concentrations | 6 month follow-up visit
  Dust will be collected from pts and assayed for indoor allergens at six months and expressed in µg/g
Fine particulate matter (PM) | 6 months
  Defined as the average PM2.5 concentration during the six month follow-up period
Use of educational material | 6 months
  Defined as the number of times educational material is downloaded from the app over the six month follow-up period
Use of the App | 6 months
  Defined as the number of visits to the app over the six month time period
Acceptability of Intervention Measure (AIM), Intervention Appropriateness Measure (IAM), and Feasibility of Intervention Measure (FIM) | 6 month follow-up visit
  4 item likert-scale validated survey, outcome will be expressed as the average score for the responses to the items at the 6 month follow-up visit. Response Scale:
  1 = Completely disagree, 2 = Disagree, 3 = Neither agree nor disagree, 4 = Agree, 5 = Completely agree. Scoring Instructions: Scales can be created for each measure by averaging responses. Scale values range from 1 to 5. No items need to be reverse coded. Higher score is a better outcome.
Number of interactions with the virtual Community Health Worker (CHW) | 6 months
  Described as the number of times pts interacted with the CHW over the six month follow up period

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Matsui, MD, Principal Investigator — University of Texas at Austin
Locations (1):
- University of Texas at Austin, Austin, Texas, United States